CLINICAL TRIAL: NCT00410527
Title: Randomized, Multi-Center, Comparative Trial of Short-Course Empiric Antibiotic Therapy Versus Standard Antibiotic Therapy for Subjects With Pulmonary Infiltrates in the Intensive Care Unit (ICU)
Brief Title: Effectiveness of Short-Course Versus Standard Antibiotic Therapy in ICU Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 999906231; 06-CC-N231
Record Dates: First submitted 2006-12-12; First posted 2006-12-13 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2007-05-22

CONDITIONS: Bacterial Infections
Keywords: Antibacterials; Colonization; Infection; Pneumonia; Resistance
MeSH Terms: conditions — Bacterial Infections; Infections; Pneumonia | interventions — Meropenem

INTERVENTIONS:
Drug: Merrem

SUMMARY:
This study will compare two treatment strategies (standard versus short-course antibiotic therapy) for preventing resistant bacterial infection in patients in the intensive care unit (ICU). ICUs are the most frequently identified source of hospital-acquired infections. This study will examine the effectiveness of 3 days of antibiotic treatment in reducing the risk of developing antimicrobial-resistant bacteria as compared with standard antibiotic therapy of at least 8 days. It will also determine whether short-course therapy can reduce the duration and costs of ICU and hospital stays, of antibiotic treatment, and of costs involving treatment of infection-related problems.

Patients of participating institutions who are in the ICU may be eligible for this study. Candidates must be 18 years of age or older. They must have been in the hospital for at least 3 days, developed new pulmonary infiltrates (fluid or cells in the airspaces of the lungs) during their ICU stay and must be at low risk of having pneumonia.

Participants on short-course therapy take antibiotic for 3 days; those receiving standard therapy take antibiotic for at least 8 days. Both groups receive the treatment intravenously (through a vein). Sputum specimens are collected at baseline (before starting therapy) and on days 3, 10, and 28. Throat culture specimens are obtained at baseline and on days 3, 10, and 28. Nasal and anal or stool samples are collected at baseline and on days 10 and 28. Cultures of respiratory specimens obtained throughout the study period are examined for evidence of antimicrobial-resistant bacteria or the isolation of a potential pathogen. All patients are followed for 28 days after enrollment or until discharge from the hospital.

DETAILED DESCRIPTION:
This study will enroll subjects who have been hospitalized at least three days (on or after fourth day of hospital stay), who have new pulmonary infiltrates during their ICU stay and who are at low risk of having pneumonia, as determined using the Clinical Pulmonary Infection Score (CPIS). The study is designed to determine whether 3 days of antibiotic treatment with meropenem (with or without coverage for MRSA) can reduce the risk of colonization with antimicrobial-resistant bacteria or the isolation of a potential pathogen compared to a standard antibiotic therapy (minimum of 8 days of therapy with antibiotics of the primary care team's choosing). The study will also examine whether short-course therapy reduces length of ICU and hospital LOS and costs based on ICU and hospital LOS, antibiotic treatment, and standardized costs related to the treatment of infection-related adverse experiences, without having a negative effect on subject mortality or the incidence of clinically significant infection.

ELIGIBILITY:
* INCLUSION CRITERIA:

The study will be limited to the medical, surgical, neurosurgical, trauma, and general ICUs of the participating institutions. Burn ICUs are not eligible for this study.

Subjects who meet all of the following criteria are eligible for enrollment into the study:

1. Subject, or legal representative, has given written informed consent.
2. Subject has developed a new pulmonary infiltrate (confirmed by radiology), after ICU admission.
3. Subject has been hospitalized at least 3 days.
4. CPIS less than or equal to 6.
5. 18 years of age or older.

EXCLUSION CRITERIA:

Subjects who meet any of the following criteria are ineligible for participation in the study:

1. Burn patients.
2. Cystic fibrosis patients.
3. Bone marrow or solid organ transplant patients.
4. Neutropenia from any cause (absolute neutrophil count (ANC) < 500), or likely to become neutropenic within 7 days.
5. Known or suspected Human Immunodeficiency Virus (HIV) infection (HIV test is not required).
6. Suspected or proven extrapulmonary infection site requiring antibiotic therapy.
7. History of anaphylaxis to penicillin or cephalosporins.
8. History of anaphylaxis to meropenem (any component of the formulation), or other carbapenems (e.g., imipenem).
9. On systemic antibiotics for more than 7 consecutive days during the previous 30 days.
10. Received more than two doses of systemic antibiotics within the past 24 hours (other than those used for surgical prophylaxis).
11. Pregnant or lactating. (Women of childbearing potential must have a negative serum or urine pregnancy test within the 7 days prior to the first dose of antibiotics.)
12. On mechanical ventilation for > 7 consecutive days during the previous 30 days.
13. Unlikely to survive past Day 7 of the study (as determined by the primary care team).
14. Previous enrollment in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0
Dates: Start 2006-08-11; Study Completion 2007-05-22

CONTACTS AND LOCATIONS:
Locations (12):
- United States (12):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Christiana Care Health Services, Newark, Delaware
  - University of Miami, Miami, Florida
  - University of Maryland, Baltimore, Baltimore, Maryland
  - Johns Hopkins Bayview Medical Center, Baltimore, Maryland
  - Baltimore VA, Baltimore, Maryland
  - Washington University School of Medicine, St Louis, Missouri
  - St. Patrick Hospital and Health Science Center, Missoula, Montana
  - Roswell Park Cancer Institute, Buffalo, New York
  - University of Oklahoma, Oklahoma City, Oklahoma
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - University of Texas, San Antonio, San Antonio, Texas

REFERENCES:
- [Background] Archibald L, Phillips L, Monnet D, McGowan JE Jr, Tenover F, Gaynes R. Antimicrobial resistance in isolates from inpatients and outpatients in the United States: increasing importance of the intensive care unit. Clin Infect Dis. 1997 Feb;24(2):211-5. doi: 10.1093/clinids/24.2.211. PMID 9114149